CLINICAL TRIAL: NCT05394298
Title: Randomized Non-inferiority Clinical Trial to Evaluate the Effectiveness and Security of Therapy for Non Complicated Enterococcal Bacteremia.
Brief Title: Short vs Long of Usual Treatment for Non Complicated Enterococcal Bacteremia
Acronym: INTENSE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Spanish Network for Research in Infectious Diseases (Other); Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT- INTENSE; 2021-003891-15 (EudraCT Number)
Record Dates: First submitted 2022-04-11; First posted 2022-05-27 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Enterococcal Bacteremia
Keywords: Enterococcus; Bacteremia
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Intervention Model Description: Randomised, multicentre, phase IV open trial of real clinical practice
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short-treatment of any active antibiotic regimen (Experimental): 7 days from the initiation of an appropriate antimicrobial therapy and documented resolution of bacteremia (negative control blood cultures performed on day 2 or 3)
  Interventions: Drug: Short-treatment of any active antibiotic regimen 7 days of any active antibiotic treatment for uncomplicated enterococcal bacteremia.
- Long-treatment of any active antibiotic regimen (Active Comparator): 14 days of any active antibiotic treatment from the date of the last positive blood culture and documented resolution of bacteremia (negative control blood cultures performed on day 2 or 3)
  Interventions: Drug: Long-treatment of any active antibiotic regimen 14 days of any active antibiotic treatment for uncomplicated enterococcal bacteremia.

INTERVENTIONS:
Drug: Short-treatment of any active antibiotic regimen 7 days of any active antibiotic treatment for uncomplicated enterococcal bacteremia. — Any active antibiotic with treatment with proven in vitro activity from a pre-stablished list of antibiotics included
  Other Names: 7 days of active antibiotics
  Arms: Short-treatment of any active antibiotic regimen
Drug: Long-treatment of any active antibiotic regimen 14 days of any active antibiotic treatment for uncomplicated enterococcal bacteremia. — Any active antibiotic with treatment with proven in vitro activity a pre-stablished list of antibiotics included
  Other Names: 14 days of active antibiotics
  Arms: Long-treatment of any active antibiotic regimen

SUMMARY:
Randomized clinical trial to determine the optimal duration of antibiotic treatment for E. Faecalis or E. faecium bacteraemia, following an innovative DOOR / RADAR (Desirability of Outcome Ranking (DOOR) and Response Adjusted for Duration of Antibiotic Risk (RADAR)) analysis methodology.

Phase IV clinical trial, open-labelled, randomized, pragmatic, multicenter study to demonstrate non-inferiority of a 7-day antibiotic regimen vs. 14 days in the treatment of bacteremia due to E. faecalis or E. faecium.

DETAILED DESCRIPTION:
Phase IV clinical trial, open-labelled, randomized, pragmatic, multicenter study to demonstrate non-inferiority of a 7-day antibiotic regimen vs. 14 days in the treatment of bacteremia due to E. faecalis or E. faecium.

Adequate antibiotic regimen is included in the protocol; initially this regimen included ciprofloxacine but this has been modified si that in the last version 3 dated feb 6th ciprofloxacine is not allowed as a possible treatment for these patients.

Antibiotic regimen included as possible treatments in the study are the follows:

* Isolated strains sensitive to ampicillin: ampicillin 2g/6 or 8h (i.v)
* Strains resistant to ampicillin and/or patients with allergy to beta-lactam drugs:
* Vancomycin: 15 mg/kg/12h i.v (with determination of trough plasma levels on day 2-3 of treatment if available).
* Linezolid: 600 mg/12 hours (i.v)
* Daptomycin: 8-10 mg/kg/day (i.v).

Intra-abdominal or soft tissue infections meeting study criteria, for which a polymicrobial infection is suspected:

Amoxicillin/clavulanic acid (isolates sensitive to ampicillin) 1 g/8h iv - Piperacillin/tazobactam (isolates sensitive to ampicillin) 4 g/8h (i.v.) - Combination of vancomycin, linezolid or daptomycin with a drug active against Gram-negative and anaerobic bacteria to ensure complete coverage in the case of bacteremia with a presumably polymicrobial focus.

Oral Treatment: In order to facilitate discharge of patients in both arms and reduce the risk of complications, as well as in keeping with the increasing use of this practice, the option to switch to oral therapy is allowed at the discretion of the responsible clinician, in both arms in patients with hemodynamic stability who tolerate oral treatment, at the discretion of the physician.

responsable.

- Amoxicillin 1g/8h or amoxicillin/clavulanic acid 875/125mg/8h if polymicrobial infection is suspected Linezolid 600mg/12h The choice will be in this order, according to the sensitivity of the isolate and allergies or other common circumstances for the use of these drugs.

The previous version allowed the use of cipro at the discretion of the clinicians as a sequential treatment option based on the fact that it is a clinical trial for low-risk bacteraemias in order to facilitate early sequential treatment (and thus avoid unnecessarily prolonging the hospital admissions.We decided to withdraw it on the basis that currently the EUCAST breakpoints only apply to urinary tract infections.The direct consequence is that the number of sequential treatment options is reduced.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or older) hospitalised with monomicrobial E. faecalis or E. faecium bacteremia.
* Negative follow-up blood cultures performed between days 2 and 3 of active treatment.
* Disappearance of fever (>37.8ºC) within the first 72 hours.
* Signed informed consent.

The previous version allowed this inclusion criterion "Early adequate control of the source of bacteremia within 72 hours in the cases in which it is feasible and necessary (urinary or biliary tract release; abscess drainage; catheter-removal, etc)", which is now removed because it is already an exclusion criterion.

Exclusion Criteria:

* patients with polymicrobial bacteremia
* Patients with limited life expectancy in whom only conservative clinical management had been decided.
* Hemodynamic instability on day 5-6 after the start of active treatment.
* Patients wearing endovascular devices or prosthetic heart valves.
* Source of uncontrolled bacteremia adequately defined as undrained abscess, bile duct infection associated with plastic prostheses not removed or not replaced within the first 72 hours of bacteraemia, other infections related to non-removed prostheses, prostatitis, and infective endocarditis, as well as infections that require prolonged treatment, such as joint and bone infections.
* Existence of a secondary focus, different from the initial one, or presence of metastatic focus of infection.
* Severe neutropenia (<500 cells / mm3) at the time of bacteremia diagnosis.
* Pregnancy and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Clinical success | TOC (Test of cure) visit (performed at day 28-32 after the end of suitable antibiotic treatment) or if drainage occurs after day 7 of treatment, TOC is to be done 7 days after that day.
  Clinical success , composite endpoint defined as all the following: (a) survival at TOC; (b) absence of enterococcal bacteremia relapse or infective endocarditis diagnosis at TOC; (c) no need to prolong therapy beyond the pre-established duration, or restart drugs against enterococci for any reason within 30 days.

SECONDARY OUTCOMES:
Rates of relapse or infective endocarditis diagnosis | TOC visit (day 28-32 ) and follow-up visit at day 90
  Rates of relapse or infective endocarditis diagnosis in the CEP (Clinically Evaluable Population)
Survival | TOC visit (day 28-32) and follow-up visit at day 90
  Number of live patients
Length of hospital stay | From patient first day inhospital (day of admission) until patient hospital discharge due to cure or home follow up assessed up to 30 days of the initiation of antibiotic administration
  Number of days patient is in-hospital
Duration of intravenous and total therapy | From date of randomization until the last follow up visit planned 30 days of the initiation of antibiotic administration
  Number of days of intravenous and total therapy in the CEP (Clinically Evaluable Population)
Incidence of diarrhoea by C. difficile | From date of randomization until the last follow up visit planned 30 days of the initiation of antibiotic administration
  To evaluate the frequency of diarrhea by C. difficile
Number of participants with Adverse Events due to antibiotic treatment | From date of randomization until the last follow up visit planned 90 days of the initiation of antibiotic administration
  Registration of all adverse events happening form the signature on informed consent form to 30 days after the study drugs administration.
Incidence of secondary infections | TOC visit (on day 28-32) and follow-up visit at day 90
  Number of patients with recurrent bacteremia
Change in SOFA score (Sepsis related Organ Failure Assessment) | Visit 0 (baseline) and TOC visit (on day 28-32) and follow-up visit at day 90
  Calculation of the SOFA score valued from 0 to 4 (0 best to 4 worst punctuation)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Eduardo López Cortés, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (22):
- Spain (22):
  - COMPLEJO Universitario de La Coruña, A Coruña, A Coruña
  - Hospital Universitario Torrecárdenas, Almería, Almeria
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - Hospital de Cruces, Barakaldo, Bizkaia
  - Hospital Universitario de Jerez de La Frontera, Jerez de la Frontera, Cadiz
  - Hospital Universitario de Puerto Real, Puerto Real, Cadiz
  - Hospital Universitario de Jaén, Jaén, JAEN
  - Hospital Universitario Costa Del Sol, Marbella, Malaga
  - Hospital Universitario Regional de Málaga, Málaga, Malaga
  - Hospital Universitario de Vigo, Vigo, Pontevedra
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Universitario Ramón y Cajal, Madrid
  - Complejo Hospitalario Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocío, Seville
  - Hospital Universitario Virgen de Valme, Seville

IPD SHARING:
Plan to Share IPD: Yes
Planning for the study will be shared with potential sites pertaining to Spanish Network for Research in Infectious Disease (REIPI)for participation. IPD is not foreseen out of this groups due to the specific characteristics of patients and sites to be candidates for study participation.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From starting to three years of study completion planification
Access Criteria: Spanish Network for Research in Infectious Disease investigators

REFERENCES:
- [Derived] Maldonado N, Rosso-Fernandez CM, Portillo-Calderon I, Borreguero Borreguero I, Tristan-Clavijo E, Palacios-Baena ZR, Salamanca E, Fernandez-Cuenca F, De-Cueto M, Stolz-Larrieu E, Rodriguez-Bano J, Lopez-Cortes LE. Randomised, open-label, non-inferiority clinical trial on the efficacy and safety of a 7-day vs 14-day course of antibiotic treatment for uncomplicated enterococcal bacteraemia: the INTENSE trial protocol. BMJ Open. 2023 Sep 6;13(9):e075699. doi: 10.1136/bmjopen-2023-075699. PMID 37673453